CLINICAL TRIAL: NCT01035294
Title: A Mindfulness-based Intervention for Treatment of Anxiety in ICD Patients
Brief Title: A Mindfulness-based Intervention for Treatment of Anxiety in ICD (Implantable Cardioverter Defibrillator) Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Elena Salmoirago-Blotcher, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-13078; 1F32AT005048-01A1 (NIH)
Record Dates: First submitted 2009-11-20; First posted 2009-12-18 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Anxiety Disorder in Conditions Classified Elsewhere

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mindfulness based intervention (Experimental)
  Interventions: Behavioral: mindfulness based intervention (MBI)
- usual care (UC) (Active Comparator)
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: mindfulness based intervention (MBI) — Eight, phone delivered, individual mindfulness sessions. Each training session will last 30 minutes (20 minutes for intervention + an additional 10 minutes for questions, answers, and for scheduling the next intervention. Patients will also receive instructions to practice at home every day, at least once a day, for at least 15 minutes. An audio CD containing guided mindfulness exercises will be given to the patient at the beginning of the study, to guide them during their home practice. The CD consists of sequences of different mindfulness techniques, consistent with the techniques learned during each session with the instructor. Each patient will record the minutes of mindfulness practice in a diary to be kept daily.
  Arms: mindfulness based intervention
Behavioral: usual care — The UC group will be offered the standard care planned by the hospital, which includes the routine care provided by the electrophysiology team and other health care professionals that the patient may see over the course of the ICD experience. All patients receive a number of printed education materials and participate to support meetings for ICD patients four times a year. Being part of the standard care offered at UMass Memorial Medical Center, these meetings are offered to all patients regardless of their assignment (thus including patients assigned to the MBI arm).
  Arms: usual care (UC)

SUMMARY:
The purpose of this study is to evaluate the feasibility and preliminary efficacy of a mindfulness-based behavioral intervention combining breathing and other relaxation exercises on symptoms of anxiety in patients undergoing the implantation of an implantable cardioverter defibrillator. This study will pilot test the feasibility and preliminary efficacy of a mindfulness-based intervention intended to improve mindfulness and anxiety levels in ICD (Implantable Cardioverter Defibrillators) patients. A randomized controlled study design will be used, in which an 8 session phone-delivered mindfulness intervention will be compared to a usual care condition among consecutive candidates for ICD procedures. The study will be conducted at the Electrophysiology (EPS) Unit at the UMass Memorial Medical Center. Assessments will be performed at baseline and at the end of the intervention (9 weeks after enrollment).

DETAILED DESCRIPTION:
The Specific Aims of this pilot study are:

Primary aim:

To determine the feasibility of a randomized clinical trial of a phone-administered, mindfulness-based training program, as measured by recruitment and retention rates, treatment adherence and fidelity.

Secondary aims:

1. To obtain preliminary estimates of the effect of a phone delivered mindfulness-based intervention on mindfulness levels, measured as the difference between baseline and post-intervention Five Factors of Mindfulness scores (FFM) in the intervention and in the control group at the end of the intervention. Hypothesis: Mindfulness levels will improve in the intervention group compared to the control group.
2. To obtain preliminary estimates of the effect of a phone delivered, mindfulness-based intervention on anxiety, measured as the difference between baseline and post-intervention Hospital Anxiety and Depression (HAD) anxiety scores in the intervention and in the control group at the end of the intervention. Hypothesis: Anxiety levels will be reduced in the intervention group, compared to the control group.
3. To collect preliminary data about the number of arrhythmic episodes/administered shocks during the intervention period. Hypothesis: the proportion of patients experiencing arrhythmic events/shocks will decrease in the intervention vs. the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21
2. ICD procedure
3. Ability to understand and speak English
4. Access to a telephone

Exclusion Criteria:

1. Inability or unwillingness to give informed consent
2. Signs of cognitive impairment (Blessed Orientation-Memory-Concentration (BOMS)scores >10)
3. New York Heart Association (NYHA) functional class>III, angina Canadian Cardiovascular Society(CCS) III and IV or clinically unstable
4. Awaiting coronary by-pass or heart transplantation
5. Co-morbid life threatening condition
6. Ongoing severe depression or psychosis

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Study feasibility | post-intervention (9 weeks after enrollment)

SECONDARY OUTCOMES:
Hospital Anxiety and Depression (HAD) anxiety scores | baseline and post-intervention (9 weeks)
Five Factors of Mindfulness scores (FFM) | baseline and post-intervention (9 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Salmoirago-Blotcher, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States